CLINICAL TRIAL: NCT02493777
Title: Ph 3 Multicenter OL Treatment-optimized RDBPC Forced-withdrawal, Parallel Grp Study to Evaluate Safety & Efficacy of Evening Dosed HLD200, a Novel DR/ER Formulation (DELEXIS) of MPH HCl in Children Aged 6-12 With ADHD in Classroom Setting
Brief Title: A Pivotal Efficacy Trial to Evaluate HLD200 in Children With ADHD in a Classroom Setting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLD200-107
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 5,10-dihydro-5-methylphenazine; Capsules; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HLD200 (methylphenidate) (Experimental): The investigational drug for this study is HLD200 MPH MR capsules comprised of the active pharmaceutical ingredient (MPH) in a dual-coated drug-layered core. Following open-label treatment optimization, subjects will be randomized (1:1) to double-blind HLD200 to be taken once daily during the evening for a period of 1-week prior to testing.
  Interventions: Drug: HLD200 methylphenidate hydrochloride (MPH) Capsules
- Placebo (Placebo Comparator): Placebo capsules will be composed of microcrystalline cellulose beads in place of MPH containing beads found in the HLD200 capsules. Following open-label treatment optimization, subjects will be randomized (1:1) to double-blind placebo to be taken once daily during the evening for a period of 1-week prior to testing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HLD200 methylphenidate hydrochloride (MPH) Capsules — HLD200 doses: 20, 40, 60, 80 or 100 mg
  Other Names: methylphenidate
  Arms: HLD200 (methylphenidate)
Drug: Placebo
  Arms: Placebo

SUMMARY:
This Phase 3 pivotal efficacy trial will examine the effects of HLD200 (methylphenidate) in patients aged 6-12 years with ADHD in a laboratory classroom setting. This study has a 6-week open-label treatment optimization period followed by a one week randomized, double-blind, placebo-controlled test phase.

DETAILED DESCRIPTION:
To address the unmet need for early morning ADHD symptom control, Ironshore has developed a novel drug delivery system that incorporates the active MPH ingredient in a delayed release/extended release formulation. This formulation provides a controlled, approximately 8-hour delay in initial drug release, followed by a subsequent controlled rate of drug release throughout the day. The goal of this system is to enable nighttime dosing of MPH to provide control of ADHD symptoms at the beginning of the next morning and throughout the remainder of the day.

The phase 3 study used an open-label treatment-optimization phase followed by a double-blind, placebo-controlled, 1-week, parallel-group treatment phase to assess safety and tolerability, as well as the time course of treatment effect, of evening-dosed HLD200 in pediatric subjects with a diagnosis of ADHD. At Visit 2, subjects began daily evening (8:00 pm ±30 minutes) treatment with 20 or 40 mg HLD200 (based on prior treatment history) for a period of 1 week and then had up to 4 additional weekly visits (Visits 3 to 6) for treatment adjustments to achieve both a) an optimal daily dose and b) an optimal treatment time prior to beginning the Double-blind Placebo-controlled Test Phase.

During Visits 3, 4, 5, and 6, investigators were permitted to titrate the dose of study drug (up or down) in 20 to 40 mg increments until either achieving the "optimal" daily dose or reaching a maximum daily dose of 100 mg/day and/or a maximum dose not exceeding 3.7 mg/kg (based on Visit 2 [baseline] weight). The final permitted dose level change was at Visit 6, after which, that dose was to be continued through Visit 7 to randomization at Visit 8. The subject underwent an assessment of study drug tolerability and, if necessary, could have his/her dose reduced. In concert with dose strength adjustments, treatment time adjustments were permitted during Visits 3, 4, 5, and 6 in increments of ±0.5 to 1.0 hour until an "optimal" treatment time was achieved (between 6:30 pm to 9:30 pm; at least 1 hour following completion of dinner). The time for changing final dose timing was at Visit 6 and continued through Visit 7 to randomization at Visit 8.

During the 1-week parallel-group phase, at Visit 8 subjects were randomly assigned (1:1 ratio) in double-blind fashion to either HLD200 or placebo treatments over the next 7 evenings. The placebo group received matching placebo at their optimal treatment time, while the HLD200 group received HLD200 at their optimal daily dose and treatment time.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be male or female children (6 to 12 years at the time of consent).
2. Subjects must have a diagnosis of ADHD as defined by DSM5 criteria and confirmation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
3. Subjects must have a Baseline ADHD-RS-IV score at or above the 90th percentile normalized for sex and age in at least 1 of the following categories: 1) Hyperactive Impulse; 2) Inattentive; or 3) Total Score. In addition, this ADHD-RS-IV Total Score must be greater or equal to 26.
4. Subjects must have a Clinical Global Impression of Severity (CGI-S) score greater than or equal to 4 and a CGI-P score >10 at the Baseline Visit.
5. Subjects who are not currently on MPH treatment must either 1) have prior experience with MPH treatment and have shown clinical response to therapy during that time; or 2) be treated with the same dose of MPH and show a clinical response with acceptable tolerability to MPH for ≥2 weeks prior to screening.
6. Parental or legal guardian confirmation of before-school function impairment and difficulties performing morning routine.
7. Regular weekday morning routine of no less than 30 minutes.
8. Subject must be considered clinically appropriate for treatment with MPH and HLD200, including ability to swallow treatment capsules.
9. Subject must be in general good health based upon medical history, physical examination, and laboratory results (including urine drug screen).
10. Subject and parent or legal guardian must be able to read, write, and/or understand at a level sufficient to provide informed consent (parent/legal guardian) and assent (subject) prior to study participation and to complete study-related materials. Subject and a parent/legal guardian must plan to be available for the entire study period.
11. Female subjects of childbearing potential (i.e., post-menarche) are required to have a negative result on urine pregnancy testing at screening (and will be given specific instructions for avoiding pregnancy during the study).
12. A medically highly effective form of birth control must be used during the study and for 90 days thereafter for subjects of either sex of childbearing potential. Examples of medically highly effective forms of birth control are as follows:

    * No sexual activity
    * Use of acceptable methods of birth control including intra-uterine device, oral, implantable, or injectable contraceptives.

Exclusion Criteria:

1. History of, or current, medical condition or laboratory result which, in the opinion of the investigator, unfavorably alters the risk-benefit of study participation, may jeopardize subject safety, or may interfere with the satisfactory completion of the study and study-related procedures.
2. Serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, or other cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
3. History of seizure disorder (except febrile seizures prior to age 5 and at least 1 year prior to study participation), Tourette's disorder, or intellectual disability of minor severity or greater (DSM5 criteria).
4. History of psychosis, bipolar disorder, anorexia nervosa, bulimia, or suicide attempt. Current depression, anxiety, conduct/behavior disorder, substance use disorder, or other psychiatric condition which, in the investigator's opinion, may jeopardize subject safety or may interfere with the satisfactory completion of the study and study-related procedures.
5. Active suicidal ideation as evidenced by an ideation score of 2 or greater on the C-SSRS.
6. History of severe allergic reaction to MPH.
7. History of no response or intolerance to the adverse effects of MPH;
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, or creatinine greater than 1.5x the upper limit of normal. Elevated bilirubin due only to Gilbert's syndrome is not exclusionary.
9. History of alcohol abuse or illicit drug use.
10. Use of prescription medications (except allowed medications; see Section 8.1.2) within 7 days of Baseline (Visit 2), except for ADHD stimulant medication (5 days) and monoamine oxidase inhibitors (MAOIs) (14 days), and over-the-counter medications (except birth control and allowed medications) within the 3 days preceding Baseline (Visit 2). Medications not covered in allowed medications or prohibited medications (Section 8.1.1) must be cleared by the medical monitor prior to enrolling the subject.
11. Participation in a clinical study with an investigational drug within the 30 days preceding study enrollment.
12. Previous treatment experience with HLD200.
13. Positive screening for illicit drug use or nicotine and/or current health conditions or use of medications that might confound the results of the study or increase risk to the subject.
14. In the opinion of the investigator, the subject may have problems complying with the protocol or the procedures of the protocol, or could face unnecessary safety risks from the study. This includes current health conditions or use of medications that might confound the results of the study or increase risk to the subject.
15. Subject's systolic or diastolic blood pressure measurement exceeds the 95th percentile for age, sex, and height at the Baseline visit.
16. Subject is significantly underweight based on Centers for Disease Control and Prevention body mass index (BMI)-for-age sex-specific values at the Screening Visit. Significantly underweight is defined as a BMI <5th percentile.
17. Subject is significantly overweight based on Centers for Disease Control and Prevention BMI-for-age sex specific values at the Screening Visit. Significantly overweight is defined as a BMI >95th percentile.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, MD, Principal Investigator — Center for Psychiatry And Behavioral Medicine Inc.
Locations (7):
- United States (7):
  - AVIDA Inc., Newport Beach, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - South Shore Psychiatric Services, PC, Marshfield, Massachusetts
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Bayou City Research, Ltd, Houston, Texas
  - Westex Clinical Investigations, Lubbock, Texas

REFERENCES:
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2025 Dec 4;12(12):CD009885. doi: 10.1002/14651858.CD009885.pub4. PMID 41342306
- [Derived] Katzman MA, Otcheretko V, Po MD, Uchida CL, Incledon B. Adverse Events During Dosing of Delayed-release/Extended-release Methylphenidate: Learnings From the Open-label Phase of a Registration Trial and a Real-world Postmarketing Surveillance Program. Clin Ther. 2023 Dec;45(12):1212-1221. doi: 10.1016/j.clinthera.2023.09.009. Epub 2023 Sep 27. PMID 37770309
- [Derived] Storebo OJ, Storm MRO, Pereira Ribeiro J, Skoog M, Groth C, Callesen HE, Schaug JP, Darling Rasmussen P, Huus CL, Zwi M, Kirubakaran R, Simonsen E, Gluud C. Methylphenidate for children and adolescents with attention deficit hyperactivity disorder (ADHD). Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD009885. doi: 10.1002/14651858.CD009885.pub3. PMID 36971690
- [Derived] Goldberg JF. Adjunctive Mood Stabilizers Are Not the Same as a Placebo-Only Arm in Bipolar Depression Trials: Reply to Terao. J Clin Psychiatry. 2021 Jun 22;82(4):21lr13919b. doi: 10.4088/JCP.21lr13919b. No abstract available. PMID 34166589
- [Derived] Terao T. Antidepressant Effects of Combined Mood Stabilizers May Account for High Placebo Response Rates. J Clin Psychiatry. 2021 Jun 22;82(4):21lr13919. doi: 10.4088/JCP.21lr13919. No abstract available. PMID 34166588
- [Derived] Childress AC, Cutler AJ, Po MD, DeSousa NJ, Warrington LE, Sallee FR, Incledon B. Symptomatic and Functional Response and Remission From the Open-Label Treatment-Optimization Phase of a Study With DR/ER-MPH in Children With ADHD. J Clin Psychiatry. 2021 Jun 22;82(4):21m13914. doi: 10.4088/JCP.21m13914. PMID 34166587
- [Derived] Childress AC, Uchida CL, Po MD, DeSousa NJ, Incledon B. A Post Hoc Comparison of Prior ADHD Medication Dose and Optimized Delayed-release and Extended-release Methylphenidate Dose in a Pivotal Phase III Trial. Clin Ther. 2020 Dec;42(12):2332-2340. doi: 10.1016/j.clinthera.2020.10.004. Epub 2020 Nov 7. PMID 33168234
- [Derived] Childress AC, Cutler AJ, Marraffino A, McDonnell MA, Turnbow JM, Brams M, DeSousa NJ, Incledon B, Sallee FR, Wigal SB. A Randomized, Double-Blind, Placebo-Controlled Study of HLD200, a Delayed-Release and Extended-Release Methylphenidate, in Children with Attention-Deficit/Hyperactivity Disorder: An Evaluation of Safety and Efficacy Throughout the Day and Across Settings. J Child Adolesc Psychopharmacol. 2020 Feb;30(1):2-14. doi: 10.1089/cap.2019.0070. Epub 2019 Aug 29. PMID 31464511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 125 participants were enrolled in this study, of which 119 were randomized to double-blind, placebo-controlled treatment at 6 sites in the United States from 28 July, 2015 to 04 March, 2015.
Pre-assignment Details: The study consisted of a screening period of up-to 4-weeks, followed by a 6-week open-label HLD200 treatment-optimization period that was followed by a 1-week randomized (1:1), placebo-controlled, double-blind period.
Groups:
- HLD200 (Methylphenidate): Participants received HLD200 capsules (containing beads with methylphenidate in a dual-coated drug-layered core; optimzed at 20, 40, 60, 80 or 100 mg) orally once daily in the evening during a 1-week randomized (1:1), placebo-controlled, double-blind-period that followed a 6-week open-label HLD200 treatment-optimization period.
- Placebo: Participants recieved placebo (matched to their dose-optimzed HLD200 capsules, but containing microcrystalline cellulose beads in place of methylphenidate) orally once daily in the evening during a 1-week randomized (1:1), placebo-controlled, double-blind period that followed a 6-week open-label HLD200 treatment-optimization period.
Period: Overall Study
Arm/Group | HLD200 (Methylphenidate) | Placebo
Started (Randomized safety population) | 65 | 54
Completed (Population completing 1-week randomized treatment) | 65 | 53
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | HLD200 (Methylphenidate) | Placebo | Total
Number analyzed (Participants) | 64 | 53 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.6 (1.58) | 9.3 (1.68) | 9.4 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 15 | 37
  Male | 42 | 38 | 80

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Kotkin, Agler, M-Flynn and Pelham Combined Score (SKAMP CS) - Model-adjusted Average of All Post-dose Time Points Assessed During a Laboratory Classroom Test Day (Visit 9).
Description: The SKAMP is a validated, 13-item, observer-rated scale designed to assess the level of impairment of classroom-observed behaviors (Wigal and Wigal, 2006). Items 1 through 4 assess subject attention; items 5 through 8 assess deportment; items 9 through 11 assess quality of work; while items 12 and 13 assess subject compliance with teacher/classroom rules. Each individual item is rated on a 7-point scale from 0 (normal, no impairment) to 6 (maximal impairment). When all individual item scores are summed together, they produce a 13-item combined score that ranges from 0 to 78, with higher scores signifying greater impairment. In the present study, the SKAMP rating scale was utilized across 9 sessions occuring at 8:00 am, 9:00 am, 10:00 am, 12:00 pm, 2:00 pm, 4:00 pm, 6:00 pm, 7:00 pm, and 8:00 pm of the laboratory classroom day. Successful training of qualified individuals on the SKAMP scale was required before raters were allowed to perform study assessments.
Time Frame: 12-hours from 8:00 am to 8:00 pm
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: SKAMP CS (12-hour average)
Arm/Group | HLD200 (Methylphenidate) | Placebo
Number analyzed (Participants) | 64 | 53
SKAMP CS (12-hour average) | 14.8 (1.17) | 20.7 (1.22)
Statistical Analysis 1: Comparison: HLD200 (Methylphenidate) vs Placebo; Test type: Superiority; p < 0.001, Mixed model repeated measures analysis

2. Secondary Outcome: Parent Rating of Evening and Morning Behavior Revised, Morning Subscale (PREMB-R AM).
Description: The PREMB-R is an 11-item rating scale designed to assess at-home functional impairments in children with ADHD during both early morning (AM) and late afternoon/evening (PM) time periods. With demonstrated validity and reliablility (Faraone et al., 2015), the AM subscale total score (sum of items 1 to 3) was designated in this study as a key secondary endpoint. Items are scored from 0 (none) to 3 (a lot), with higher scores signifying greater impairment of function. The PREMB-R rating scale was completed by parents during the 2-days prior to study visits at the beginning and end of the open-label period (Visits 2 and 8, respectively), as well as at the end of the randomized, double-blind period (Visit 9). At each visit, these ratings were used only for review by the clinician (MD, PhD, DO, licensed social worker, or any trained mental health professional approved by the sponsor) as part of a structured interview to enable collection of a clinician-rated PREMB-R AM subscale score.
Time Frame: PREMB-R AM mean subscale score for the 2-days prior to Visit 9.
Population: Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: PREMB-R AM subscale total score
Arm/Group | HLD200 (Methylphenidate) | Placebo
Number analyzed (Participants) | 64 | 53
PREMB-R AM subscale total score | 0.9 (0.27) | 2.7 (0.27)
Statistical Analysis 1: Comparison: HLD200 (Methylphenidate) vs Placebo; Test type: Superiority; p < 0.001, Mixed model repeated measures analysis

ADVERSE EVENTS:
Time Frame: Adverse events were collected across the duration of the study (up to 13-weeks). However, an adverse event is considered treatment-emergent during the randomized, placebo-controlled phase only if it started on or after the first dose of double-blind study medication, but before the last dose of double blind study medication plus 72 hours as reflected in the table below.
Description: Adverse events were recorded by study staff at every post-screening study visit based on spontaneous report from subjects/parents, regardless of causality. However, sleep-related adverse event were directly solicited from subjects/parents by study staff using a structured interview format to assessing sleep disturbances (e.g., issues with sleep onset, quality and quantity), rather than obtained from spontaneous reporting.
Arm/Group | HLD200 (Methylphenidate) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/54
Other Adverse Events (participants affected / at risk) | 14/65 | 12/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HLD200 (Methylphenidate) (N=65) | Placebo (N=54)
Any Insomnia (Psychiatric disorders) | 5 | 5 — Any Insomnia is a combined sleep-related AE term which includes Initial, Middle and Terminal insomnias (Note: There were no reported adverse events of the Insomnia, not specified term during the double blind period.
Blood pressure diastolic increased (Investigations) | 9 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes